CLINICAL TRIAL: NCT01229995
Title: A Comparison of Zirconia CAD/CAM and Conventionally Fabricated Single Implant Abutments and Restorations in the Esthetic Zone: a Randomized Controlled Clinical Trial.
Brief Title: Randomized Controlled Clinical Trial of CAD/CAM and Conventionally Fabricated Singl Implant Abutments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: German O. Gallucci, Harvard School of Dental Medicine
Allocation: Randomized
Other Study IDs: M17719-104
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Missing Teeth; Teeth Replacemnt by Single Dental Implant; Zirconia Abutment; Titanium Abutment
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prefabricated Abutment (Active Comparator)
  Interventions: Device: dental implants - zirconia abutmetns - prefabricated abutments

INTERVENTIONS:
Device: dental implants - zirconia abutmetns - prefabricated abutments

SUMMARY:
CAD/CAM technology has been introduced to the field of implant dentistry in the beginning of 1990's (Priest 2005). Since their introduction, the use of CAD/CAM technology in the production of dental implant restorations has been rapidly expanding. However, little evidence is currently present supporting its clinical viability (Henriksson 2003, Canullo 2007).

Therefore, the suggested prospective randomized study includes bone level placed Straumann implants restored with transmucosal elements and crowns fabricated using either CAD/CAM "Etkon" technology (Zirconia abutment and ceramic crown) or a conventional technique (Crossfit titanium abutment and a ceramometal crown).

The aim of this randomized controlled clinical trial is to examine single-tooth implant restorations in the esthetic zone. An esthetic area is defined as any area that is visible in the patient's full smile. [3rd ITI consensus conference 2004] The rehabilitations will be fabricated using two different techniques. Zirconia CAD/CAM (ZCC) implant restorations (tests) will be compared to Titanium conventionally-fabricated (TCF) implant restorations (controls) using, reproducible esthetic (objective/subjective) and biologic parameters.

This in vivo study is a randomized study with two groups of 15 patients with one implant each for a total of 30 patients and 30 implants. The implants will be examined for successful tissue integration according to the criteria of success (Buser et al. 1990) at every recall visit.

In addition, the following parameters will be evaluated for each restoration:

* Esthetic: A. Objective: PES/WES Score (Belser et al. 2009) from 1:1 digital photograph, study casts, and spectrophotometric measurements, and B. Subjective: VAS questionnaire for patients and VAS questionnaire from experts.
* Biologic (mPI, mB, simplified GI, microbial sample, periapical radiograph for DIB, and width of keratinized facial mucosa)

Finally, an evaluation of the mechanical, biologic and technical complications will be performed at every recall visit. Mechanical complications would be defined as those complications that involve the prosthesis such as abutment screw loosening, fracture of the veneer material, fracture of the crown framework, abutment screw fractures, and implant fractures. The category of biologic complications will include those complications that involve the soft tissues (e.g., fistula, suppuration, bleeding, gingival inflammation, and soft tissue dehiscence). Technical complications are defined as those related to restorative components and crowns (e.g. crown emergence profile, abutment and crown fit, screw loosening, ceramic fracture).

DETAILED DESCRIPTION:
Introduction

Long-term prospective studies demonstrate a high success rate of Straumann implants in partially or fully edentulous patients both with early and conventional loading (Salvi et al. 2004, Lambrecht et al. 2003, Cochran et al. 2002, Weber et al. 2000, Buser et al. 1997). Before the introduction of CAD/CAM technology to the field of implant dentistry in the beginning of 1990's (Priest 2005), the available approach for restoring single dental implants was either with stock or cast custom abutments and a ceramo-metal crowns. In spite of the satisfactory results that this conventional treatment approach has achieved, several disadvantages have been recognized. First, non tooth-colored abutments possess the problem of bluish appearance of overlying tissue in cases of thin gingival biotype (Barclay et al. 1996, Prestipino and Ingber, 1996). Second, with stock abutments ideal emergence profile can not be achieved (Daftary 1997), a disadvantage that was reduced with the use of custom abutments. However, custom abutments present other disadvantages including possible imprecision of fit due to inaccuracies associated with impression, waxing, investing and casting procedures and the negative effect of the gold alloy on the peri-implant mucosal barrier as demonstrated by Abrahamsson in 1998 (Abrahamsson et al 1998 ).

The introduction of CAD/CAM technology to implant dentistry was meant to provide higher quality restorations. Since its introduction, the use of this technology in the production of implant ceramic frameworks and crowns especially in esthetic regions has been rapidly expanding because of the promising esthetic, biologic, and mechanical properties. Alumina as well as Zirconia abutments are characterized by good tissue compatibility (Abrahamsson et al. 1998). In a study by Barclay et al in 1996 it was found that plaque accumulation scores for ceramic-coated transmucosal elements were significantly lower than those recorded in titanium transmucosal elements (Barclay et al. 1996). These results suggest that the further development of a ceramic implant transmucosal collar may assist plaque control at the soft tissue-implant interface and may favorably influence the tissues in this region (Barclay et al. 1996). Other studies documented no significant differences in plaque accumulation and microbial colonization between titanium and ceramic abutment samples (Andersson et al. 2003, Rasperini et al. 1998). The bacterial colonization of Zirconia ceramic surfaces was recently studied in vitro and in vivo (Rimondini et al. 2002). The authors found that, overall, Zirconia ceramic surfaces developed for implant abutments accumulate fewer bacteria than commercially pure titanium, and may therefore be considered as a promising material for abutment manufacturing (Rimondini et al. 2002). A comparison of the recorded superficial soft tissue responses to titanium and ceramic surfaces of transmucosal elements of implants revealed no significant differences between both groups (Barclay et al. 1996, Andersson et al. 2001). Almost no marginal bone loss was recorded, indicating a stable bone situation both at ceramic and titatium abutments on single-tooth implants (Andersson et al. 2001). However, it seems to be that the peri-implant soft tissues adjacent to titanium and ceramic surfaces may differ in features that are not apparent when routine clinical parameters are used (Barclay et al. 1996).

Because of their specific mechanical properties, all-ceramic restorations demonstrate a lower fracture resistance than ceramic restorations supported by metal substructures. The ceramic abutments on implants are more sensitive to fracture and to handling procedures than the titanium abutments (Andersson et al. 2001). However, advances have been made in the fabrication of high-strength all-ceramic abutments for anterior implants (Yildirim et al. 2003). The hardness of the Zirconium ceramic also allows it to undergo conventional prophylaxis with ultrasonic scalers without alteration of its surface quality of abutment (Marzouk, 1996). Moreover, Zirconia has a flexural strength and fracture toughness almost twice as high as alumina (Glauser et al. 2004, Yildirim et al. 2003).

Currently very limited number of clinical studies is present supporting the clinical viability of CAD/CAM ceramic restorations (Henriksson 2003, Canullo 2007) and no reports were found on the performance of CAD/CAM ceramic implant restorations in comparison to conventional implant restorations.

Objective:

The aim of this randomized controlled clinical trial is to examine single-tooth implant abutments and restorations in the esthetic zone. Restorations will be fabricated using two different techniques. Zirconia CAD/CAM (ZCC) implant abutments and restorations will be compared to conventional, prefabricated Titanium (TCF) implant abutments and porcelain-fused-to-metal restorations using reproducible aesthetic (objective/subjective) and biologic parameters.

Hypothesis:

The hypothesis of this investigation is that ZCC implant abutments/restorations (test group) will achieve better biologic and esthetic outcomes when compared with TCF types (control group). The null hypothesis is defined as follows: ZCC implant abutments/restorations and TCF implant restorations are indistinguishable when biologic and esthetic outcomes are compared.

Clinical Significance:

CAD/CAM technology has been involved in the fabrication of dental abutments and restoration for the purpose of improving the biologic and esthetic results. This assumption has been formulated primarily from subjective interpretations as objective assessments from randomized controlled trials are sparse at best. This study will be significant for clinical dentistry in that it will create evidence on the clinical long-term performance of Zirconium CAD/CAM abutments and ceramic crowns compared to stock titanium abutments and porcelain-fused-to-metal restorations using subjective and objective evaluation parameters that will be statistically compared.

Materials and Methods:

Patients with an indication for an implant supported single tooth restoration in the esthetic zone will be included in the study according to the following criteria:

Inclusion Criteria:

General:

1. Age > 21 years
2. Absence of relevant medical conditions
3. Absence of periodontal diseases
4. The opposing dentition must be natural teeth or fixed (not removable) restorations on teeth or implants.
5. Availability for 5-year follow-up

Local:

1. One missing tooth in the esthetic zone. An esthetic area is defined as any area that is visible in the patient's full smile. [3rd ITI consensus conference 2004]
2. Presence of two intact adjacent teeth which are either non-restored or with minor restorations (small composite restorations)
3. Adequate native bone to achieve primary stability
4. Adequate band of keratinized mucosa (at least 2mm)
5. Full Mouth Plaque Scores (FMPS) and Full Mouth Bleeding Scores (FMBS) < 25 %

Exclusion criteria

General:

1. Heavy smokers (more than 10 cigarettes/day)
2. Presence of conditions requiring chronic prophylactic use of antibiotics
3. Medical conditions requiring prolonged use of steroids.
4. History of radiation therapy to the head or neck or history of chemotherapy.
5. Physical handicaps that would interfere with the ability to perform adequate oral hygiene.
6. Patients with inadequate oral hygiene.

Local:

1. Adjacent implant
2. Presence of periapical radiolucencies at the adjacent teeth
3. Missing adjacent teeth
4. Local inflammation, including untreated periodontitis.
5. Persistent intraoral infections.
6. Untreated mucosal diseases.

Subject population Patients will be recruited from the patient pool of the Teaching and Faculty Practice at the Harvard School of Dental Medicine. A 12-month period will be allowed to enroll the patients in this study. The mean treatment outcome will be compared between the two randomized patient groups, allowing for detection of the smallest clinically important differences between these means (TheSealedEnvelope™- http://www.thesealedenvelope.com/ power.php).

Patient entry (informed consent, patient registration, randomization and blinding) An informed consent approved by the Harvard Medical School/Harvard School of Dental Medicine Committee on Human Studies will be obtained for all subjects to be entered in this study. Its conduct will adhere to the principles outlined by the Office for Research Subject Protection of the Harvard Medical School / Harvard School of Dental Medicine. Each subject will be randomly assigned to one of the two treatment options. A random permuted block approach will be used to allocate patients into one of the treatment groups. A sealed envelope containing the treatment group (control or test group) will be assigned to each patient. Subsequently and according to the assigned treatment, a ZCC restoration (test group) or a TCF ceramo-metal (control group) will be fabricated and delivered to the clinician.

For subjective evaluation the trial design will be on a double blinding level, which means that neither patients nor expert clinicians will know which treatment the patients are randomized to. This can be achieved by concealing allocation information from patients and by using expert clinicians, who are otherwise not involved in the patients' care, to assess treatment difficulties and outcomes without knowing their treatment group.

Treatment groups

30 patients will be randomly allocated to control or test group presented in Table (1)

Group (n= 30 patients) Implant Abutment Crown Loading Test group (n=15) ZCC BL Straumann Etkon Zirconia Cement-retained Etkon Zirconia 6-8 weeks control group (n=15) TCF BL Straumann Crossfit titanium Cement-retained PFM 6-8 weeks

Evaluation Parameters and time schedule:

Patients will be evaluated for esthetic (objective and subjective parameters) and biologic parameters as well as the success criteria through out the study period. The baseline measurements are defined as the measurements taken during the healing period after insertion of bone level implant.

During the healing period, after insertion of a Straumann Bone Level implant following standard surgical procedures, patients will use removable provisional prostheses.

The implants will be examined for successful tissue integration according to the criteria of success (Buser et al. 1990) at every recall.

Criteria of success:

1. Absence of persistent subjective complaints, such as pain, foreign body sensation and/or dysaesthesia
2. Absence of a recurrent peri-implant infection with suppuration
3. Absence of mobility
4. Absence of a continuous radiolucency around the implant

Esthetic parameters :

Objective parameters

* Standardized intra-oral digital photograph (1:1 magnification) An intra-oral photograph will be taken, positioning the plane of the camera body parallel to the vestibular face of the teeth adjacent to the single edentulous gap. (Figure 1)
* Papilla Height: Distance between the mesial and distal papilla and the zenith of the mid-facial gingival margin of the adjacent teeth The distance from the most coronal part of the mesial and distal papillae to the zenith of adjacent teeth, will be measured from study casts and digital photographs. (Figure 2)
* Buccal gingival margin measurement: Distance between the mid-facial gingival margin and the incisal edge of adjacent teeth The distance from the zenith of adjacent teeth to the most coronal part of the incisal edge, will be measured from study casts and digital photographs. This measurement will serve to determine the buccal gingival recession/growth when compared with further measurements. It will be recorded as "0" at baseline. (Figure 3)
* Study cast
* Spectrophotometer recording at adjacent teeth. A spectrophotometer (Crystaleye, Olympus, Japan) will be used to select and digitally record the shade for each adjacent tooth. The sterilizable adapter of the spectrophotometer's intra-oral camera will be positioned on the alveolar process over the respective adjacent tooth. Once the resulting video image of the tooth is centered in an orthoradial way in the measuring square depicted on the computer screen, the spectrophotometric data will be recorded three consecutive times for each tooth. This data will be later compared with records obtained from final crowns by repeating the spectrophotometer measurement over the control and test group restorations. (Figure 4)
* Buccal periimplant mucosa margin: Distance between mid-facial gingival margin and incisal edge of the implant restoration At implant crown insertion, the distance from the zenith of the implant restoration to the most coronal part of the incisal edge will be measured from study casts and digital photographs. This measurement will serve to determine the buccal gingival recession/growth when compared with further measurements. It will be recorded as "0" at the implant crown insertion. (Figure 5)

Subjective parameters:

1. Visual Analogue Scale (VAS) of patient's judgment on:

   * At baseline: detriment of his/her esthetic appearance and respective expectations
   * At crown insertion:

     * Overall treatment satisfaction
     * Accomplishment of initial expectations
   * At 1, 6 months, 1, 3 and 5 year follow up:

     * • Overall treatment satisfaction
     * • Impact on self-esteem
     * • Functionality
2. Visual Analogue Scale (VAS) of 3 expert clinicians' judgments on the case difficulty

Parameters Follow-up time schedule Baseline At insertion 1 month 6 months 1 year 3 years 5 years

Esthetic:

Objective:

1. 1:1 digital photograph
2. Papilla height
3. Buccal gingival margin
4. Study cast
5. Spectrophotometer
6. Buccal periimplant mucosa margin

Subjective:

1. (VAS) questionnaire for patients
2. (VAS)questionnaire from experts

Biologic parameters

1. mPI Modified plaque index (Mombelli et al. 1987) for evaluation of oral hygiene standard: 0: No detection of plaque; 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant; 2: Plaque can be seen by the naked eye; 3: Abundance of soft material.
2. mBI Modified sulcus bleeding index (mBI) (Mombelli et al. 1987): 0: No bleeding when a periodontal probe is passed a long the gingival margin adjacent to the implant; 1: Isolated bleeding spots visible; 2: Blood forms a confluent red line on margin; 3: Heavy or profuse bleeding.
3. simplified GI Simplified Gingival Index (Apse et al. 1991): 0: Normal mucosa; 1: Minimal inflammation with color change and minor edema; 2: Moderate inflammation with redness, edema and glazing; 3: Severe inflammation wit redness, edema, ulceration and spontaneous bleeding without probing.
4. Microbiological sample Microbial samples from a tooth in the same sextant as the implant and from the implant healing cap prior to its initial removal at the start of the restorative procedures will be obtained. Additional samples will be taken at 1month, 6, 12, 36 and 60 months after the insertion of the restoration. The samples will be analysed for P. gingivalis, T. forsythia (B. forsythus) T..denticola, .F. nucleatum, P. micra (P. micros) P. nigrescens, P. intermedia, C. rectus, C. gracilis, E. nodatum and S. constellatus. (Quirynen et al. 2002, Keller et al. 1998, Conrad et al. 1996). Sample analysis will be performed at the Forsyth Institute, Boston, MA, on a contractual basis. Samples will be identified only by their number for this purpose. No patient identifying data will be revealed. The correlation between the periimplant microflora before and after loading within the same subject as well as potential differences in quantity and composition of the microflora of ZCC and TCF implant abutments and restorations will be analysed.
5. Standardized periapical radiograph to assess DIB values. Standardized peri-apical long cone parallel radiographs of the implant (Harris et al. 2002) will be taken. For standardization of radiographs, a film holder will be attached to a custom-made bite splint. This same device will be used during the whole study for radiographic records. From these radiographs, bone resorption will be measured as distance from the implant shoulder to first bone-to-implant contact (DIB). (Figure 6)
6. Width of keratinized facial mucosa

Parameters Follow-up Time schedule Baseline Crown Insertion 1 mos 6 mos 1 year 3 years 5 years

Biologic:

1. mPI (modified Plaque Index)
2. mBI (modified sulcus Bleeding Index)
3. simplified GI (Gingival Index)
4. microbiological sample
5. PA (Periapical X-ray for DIB)
6. Width of keratinized facial mucosa

D. Mechanical, Biologic and Technical complications An evaluation of the mechanical, biologic and technical complications will be performed at every recall visit. Mechanical complications would be defined as all those complications that involve the prosthesis such as abutment screw loosening, fracture of the veneer material, fracture of the crown framework, abutment screw fractures, and implant fractures. The category of biologic complications will include the complications that involve the soft tissues ex. fistulas, suppuration, bleeding, gingival inflammation, and soft tissue dehiscence. Technical complications would be defined as those complications that are related to lab procedures and fabricating techniques ex. abutment and crown emergence profile, abutment and crown fit.

Complications Follow-up Time Schedule Baseline At insertion 1 mo 6 mos 1 year 3 years 5 years

Mechanical:

1. Abutment screw loosening
2. Fracture of a veneer material
3. Fracture of the crown framework
4. Fractures of abutment screws
5. Fractures implants

Biologic:

1. Fistulas
2. Suppuration
3. Bleeding
4. Gingival inflammation
5. Soft tissue dehiscence

Technical:

1. Abutment emergence profile
2. Crown emergence profile
3. Abutment fit
4. Crown fit

Statistical Analysis: After data collection and completion of the investigation, a one-way analysis of variance (ANOVA) will be used to compare the mean values of all objective and subjective parameters. Their variance will be broken down into two components: (a) "between groups" component (control group vs. test group) at baseline, crown insertion, and each follow-up period and (b) "within group" component at baseline, crown insertion, and each follow-up period. A multiple LSD range test (confidence level 95%) will be applied to determine which means differ statistically from each other.

Timetable June 2009 beginning of the study May 2010 deadline for patients' entry and allocation August 2010 deadline for data collection of baseline and crown insertion measurements September 2010 deadline for data collection of 1-month follow up measurements February 2011 deadline for data collection of 6-month follow up measurements August 2011 deadline for data collection of 12-month follow up measurements August 2012 deadline for data collection of 24-month follow up measurements August 2013 deadline for data collection of 36-month follow up measurements August 2014 deadline for data collection of 48th month follow up measurements August 2015 deadline for data collection of 60th month follow up measurements February 2016 deadline for final publication of data

References

* Abrahamsson I, Berglundh T, Glantz PO, Lindhe J. The mucosal attachment at different abutments. An experimental study in dogs. J Clin Periodontol. 1998;25(9):721-7.
* Andersson B, Glauser R, Maglione M, Taylor A. Ceramic implant abutments for short-span FPDs: a prospective 5-year multicenter study. Int J Prosthodont. 2003;16(6):640-6.
* Andersson B, Taylor A, Lang BR, Scheller H, Scharer P, Sorensen JA, Tarnow D. Alumina ceramic implant abutments used for single-tooth replacement: a prospective 1- to 3-year multicenter study. Int J Prosthodont. 2001;14(5):432-8.
* Barclay CW, Last KS, Williams R. The clinical assessment of a ceramic-coated transmucosal dental implant collar. Int J Prosthodont. 1996;9(5):466-72.

Belser UC, Gruetter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth Implants using objective esthetic criteria:

a cross-sectional retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol 2009; 80: 140-151.

* Buser D, Mericske-Stern R, Bernard JP, Behnecke A, Behnecke N, Hirt HP; Belser UC, Lang NP. Long-term evaluation of non-submerged ITI implants. Part 1: 8-year life table analysis of a prospective multi-center study with 2359 implants. Clin Oral Implants Res. 1997;8(3):161-72.
* Canullo, L., Clinical outcome study of customized zirconia abutments for single-implant restorations. Int J Prosthodont, 2007. 20(5): p. 489-93.
* Cochran DL, Buser D, ten Bruggenkate CM, Weingart D, Taylor TM, Bernard JP, Peters F, Simpson JP.The use of reduced healing times on ITI implants with a sandblasted and acid-etched (SLA) surface: early results from clinical trials on ITI SLA implants. Clin Oral Implants Res. 2002;13(2):144-53.
* Daftary F. Dentoalveolar morphology: evaluation of natural root form versus cylindrical implant fixtures. Pract Periodont aesthet Dent. 1997; 9:469.
* Glauser R, Sailer I, Wohlwend A, Studer S, Schibli M, Scharer P. Experimental zirconia abutments for implant-supported single-tooth restorations in esthetically demanding regions: 4-year results of a prospective clinical study. Int J Prosthodont. 2004;17(3):285-90.
* Henriksson, K. and T. Jemt, Evaluation of custom-made procera ceramic abutments for single-implant tooth replacement: a prospective 1-year follow-up study. Int J Prosthodont, 2003. 16(6): p. 626-30.
* Lambrecht JT, Filippi A, Kunzel AR, Schiel HJ. Long-term evaluation of submerged and nonsubmerged ITI solid-screw titanium implants: a 10-year life table analysis of 468 implants. Int J Oral Maxillofac Implants. 2003;18(6):826-34.
* Marzouk J. Two applications of transmucosal milled ceramic in implantology: preliminary clinical examples. Quintessence Int. 1996;27(8):533-47.
* Prestipino V, Ingber A. All-ceramic implant abutments: esthetic indications. J Esthet Dent. 1996;8(6):255-62.
* Priest G. Virtual-designed and computer-milled implant abutments. J Oral Maxillofac Surg. 2005; 63:22-32.
* Rasperini G, Maglione M, Cocconcelli P, Simion M. In vivo early plaque formation on pure titanium and ceramic abutments: a comparative microbiological and SEM analysis. Clin Oral Implants Res. 1998;9(6):357-64.
* Rimondini L, Cerroni L, Carrassi A, Torricelli P. Bacterial colonization of zirconia ceramic surfaces: an in vitro and in vivo study. Int J Oral Maxillofac Implants. 2002;17(6):793-8.
* Salvi GE, Gallini G, Lang NP. Early loading (2 or 6 weeks) of sandblasted and acid-etched (SLA) ITI implants in the posterior mandible. A 1-year randomized controlled clinical trial. Clin Oral Implants Res. 2004;15(2):142-9.
* Weber HP, Crohin CC, Fiorellini JP. A 5-year prospective clinical and radiographic study of non-submerged dental implants. Clin Oral Implants Res. 2000;11(2):144-53.
* Yildirim M, Fischer H, Marx R, Edelhoff D. In vivo fracture resistance of implant-supported all-ceramic restorations. J Prosthet Dent. 2003;90(4):325-31.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

General:

1. Age > 21 years
2. Absence of relevant medical conditions
3. Absence of periodontal diseases
4. The opposing dentition must be natural teeth or fixed (not removable) restorations on teeth or implants.
5. Availability for 5-year follow-up

Local:

1. One missing tooth in the esthetic zone. An esthetic area is defined as any area that is visible in the patient's full smile. [3rd ITI consensus conference 2004]
2. Presence of two intact adjacent teeth which are either non-restored or with minor restorations (small composite restorations)
3. Adequate native bone to achieve primary stability
4. Adequate band of keratinized mucosa (at least 2mm)
5. Full Mouth Plaque Scores (FMPS) and Full Mouth Bleeding Scores (FMBS) < 25 %

Exclusion Criteria:

Exclusion criteria

General:

1. Heavy smokers (more than 10 cigarettes/day)
2. Presence of conditions requiring chronic prophylactic use of antibiotics
3. Medical conditions requiring prolonged use of steroids.
4. History of radiation therapy to the head or neck or history of chemotherapy.
5. Physical handicaps that would interfere with the ability to perform adequate oral hygiene.
6. Patients with inadequate oral hygiene.

Local:

1. Adjacent implant 2. Presence of periapical radiolucencies at the adjacent teeth 3. Missing adjacent teeth 4. Local inflammation, including untreated periodontitis. 5. Persistent intraoral infections. 6. Untreated mucosal diseases.

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05

PRIMARY OUTCOMES:
The aim of this randomized controlled clinical trial is to examine single-tooth implant abutments and restorations in the esthetic zone.

SECONDARY OUTCOMES:
Test group will achieve better biologic and esthetic outcomes when compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: German O. Gallucci, DMD Dr.Med.Dent., Principal Investigator — Harvard School of Dental Medicine